CLINICAL TRIAL: NCT04018209
Title: Aquagenic Pruritus in Myeloproliferative Neoplasms
Acronym: PANAM
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: PANAM (29BRC19.0001)
Record Dates: First submitted 2019-05-24; First posted 2019-07-12 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Deciphering Aquagenic Pruritus in Myeloproliferaitive Neoplasms
Keywords: Pruritus; Myeloproliferative Neoplasms
MeSH Terms: conditions — Pruritus; Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Description of the characteristics of aquagenic pruritus expressed by patients suffering from myeloproliferative neoplasms.

Prospective work based on the distribution of a dedicated questionnaire.

DETAILED DESCRIPTION:
Patients with myeloproliferative neoplasms identified and followed in French Hospitals. Patients could be followed for polycythemia vera or essential thrombocythemia or primary myelofibrosis.

Distribution of the questionnaire to each patient with myeloproliferative neoplasm (treated or not) suffering from aquagenic pruritus.

Analyse of each characteristic of the aquagenic pruritus by a statistician and publication at the end.

ELIGIBILITY:
Inclusion Criteria:

* Patients with one of three non-chromosomal Philadelphia-positive myeloproliferative neoplasms: polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF).
* Suffering (or having suffered) from aquagenic pruritus.
* No age limit, but major
* Patient having formulated his non-opposition

Exclusion Criteria:

* Patients with MPN with non-aquagenic pruritus,
* Patients with another hematologic disease and aquagenic pruritus
* Patients unable to complete the questionnaire.
* Patients with physical or mental disabilities to formulate non-opposition
* Refusal of participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with one of three Philadelphia positive non-chromosome myeloproliferative neoplasms: polycythemia vera (PV), essential thrombocythemia (TE) or primary myelofibrosis (PMF).
  And suffering (or having suffered) from aquagenic pruritus.
Sampling Method: Probability Sample
Enrollment: 170 (Actual)
Dates: Start 2019-07-09 (Actual); Primary Completion 2020-01-09 (Actual); Study Completion 2021-01-06 (Actual)

PRIMARY OUTCOMES:
Description of pruritus in patients with myeloproliferative neoplasms | at the time of questionnaire completion (Day 0)
  Intensity of pruritus (visual analogic scale)

SECONDARY OUTCOMES:
Description of therapies used to treat pruritus | at the time of questionnaire completion (Day 0)
  Name of drugs used

CONTACTS AND LOCATIONS:
Locations (11):
- France (11):
  - 05, Lyon, Auvergne Rhônes-alpes
  - 10, Quimper, Brestagne
  - 11, Morlaix, Brittany Region
  - 09, Saint-Brieuc, Brittany Region
  - 07, Saint-Louis, Grand Est
  - 03, Annecy, Haute-Savoie
  - 04, Roubaix, Hauts-de-France
  - 08, Rochefort, Nouvelle-Aquitaine
  - 06, Angers, Pays de la Loire Region
  - 02, Villejuif, Val-de-marne
  - 01, Brest

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning six months and ending five years following the publication
Access Criteria: Data access requests will be rewiewed by internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.